CLINICAL TRIAL: NCT02677220
Title: Implantation With the Nucleus CI532 Cochlear Implant in Adults
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: No enrolled subjects
Sponsor: Cochlear (Industry)
Collaborators: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAM5631; NCT02560987 (obsolete NCT alias)
Record Dates: First submitted 2016-02-03; First posted 2016-02-09 (Estimated); Results first posted 2019-03-12 (Actual); Last update posted 2019-03-12 (Actual); Status verified 2019-02

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Surgical (Experimental): Subjects to be implanted with the CI532 cochlear implant in one ear
  Interventions: Device: CI532 cochlear implant

INTERVENTIONS:
Device: CI532 cochlear implant

SUMMARY:
The aim of this study is to investigate the clinical benefit for patients implanted with the Nucleus® CI532 cochlear implant.

The Nucleus® CI532 has a pre-curved, perimodiolar array, the EA32, which is introduced into the cochlea through a straightening sheath.

ELIGIBILITY:
Inclusion Criteria:

* Meet current cochlear implant criteria at the implanting center
* 18 years or older with bilateral sensorineural hearing loss
* Limited benefit from appropriate binaural hearing aids
* Moderate to profound hearing loss in the low frequencies and profound hearing loss in the mid to high frequencies
* Preoperative unaided threshold between 40 and 65 dB HL, inclusively, at 250 Hertz (Hz) and 500 Hz in the ear to be implanted
* Fluent speaker in the language used to assess clinical performance

Exclusion Criteria:

* Evidence of hearing loss prior to age 5
* Sensorineural severe to profound hearing loss greater than 20 years at and above 2000Hz
* Simultaneous bilateral implantation prior to the study
* Medical or psychological conditions that contraindicate undergoing general anesthesia or surgery
* Cochlear anomaly that might prevent complete insertion of the electrode array
* Hearing impairment due to lesion or neuropathy of the acoustic nerve, VIII nerve, or central auditory pathway
* Active middle ear infection
* Tympanic membrane perforation
* Unrealistic expectations
* Unwillingness or inability co comply with all investigational requirements
* Patients with existing cerebral shunts or drains
* Recurrent episodes of bacterial meningitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2016-05-11 (Actual); Primary Completion 2017-08-23 (Actual); Study Completion 2017-08-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- NYU Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Surgical: Subjects implanted with the CI532 cochlear implant in one ear
Period: Overall Study
Arm/Group | Surgical
Started | 1
Completed | 0
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Surgical
Number analyzed (Participants) | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: AzBio Sentence Recognition in Noise
Description: The AzBio Sentence test was recorded at 3 months prior to subject withdraw. Not collected at endpoint. AzBio Tests consists of 15 lists of 20 sentences each. AzBio sentences are spoken by different talkers in a conversational style with limited contextual cues that the listener can use to predict or 'fill in' unintelligible words. Each list includes 5 sentences from 4 different male and female speakers. Each word in the sentence counts toward the overall score and the resulting score is presented in percent correct.
Time Frame: 3 months post-activation
Measure: Mean (Standard Deviation); unit: percent correct
Arm/Group | Surgical
Number analyzed (Participants) | 1
percent correct | 35 (0)

2. Secondary Outcome: Glasgow Benefit Inventory
Description: The Glasgow Benefit Inventory (GBI) is a health utility assessment used at six months post-operatively. Performance benefits are a change in score from pre- to post-operatively, scored from -100 to +100.
Time Frame: 6 months post-activation
Population: subject did not reach endpoint - GBI was not collected at 3 months per protocol
Arm/Group | Surgical
Number analyzed (Participants) | 0

3. Secondary Outcome: Speech, Spatial, and Qualities of Hearing Scale
Description: The Speech Spatial and Qualities of Hearing Scale (SSQ) is a subjective measure of satisfaction. Change is reflected in a gain in scores pre- to post-operatively (-10 to +10).
Time Frame: 6 months post-activation
Population: subject did not reach endpoint - SSQ was not collected at 3 months per protocol
Groups:
- Surgical: Subjects with the CI532 cochlear implant in one ear
Arm/Group | Surgical
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 8 months
Description: SAE October 2016 - blood and pus draining from the incision. Antibiotics prescribed.
  November 2016 - resolved. Initial activation of the device. December 2016 through April 26, 2017 - continued drainage and treatment using a combination of routine wound care and oral antibiotics.
  June 2017 - Explantation required July 2017 - Withdrawn - test device was no longer in place.
Arm/Group | Surgical
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 1/1
Other Adverse Events (participants affected / at risk) | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Surgical (N=1)
Device Explant (Ear and labyrinth disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2016-04-16): https://cdn.clinicaltrials.gov/large-docs/20/NCT02677220/Prot_000.pdf